CLINICAL TRIAL: NCT05722457
Title: Comparison of the Effects of External Focus and Internal Focus Instructions Applied in Balance Training on Individuals With Chronic Low Back Pain: Randomized Controlled Trial
Brief Title: Comparison of the Effects of External Focus and Internal Focus Instructions Applied Chronic Low Back Pain: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Safak Kuzu, Research Assistant/Araştırma Görevlisi, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-0003-0145-3565
Record Dates: First submitted 2022-12-30; First posted 2023-02-10 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Physical Therapy Techniques
Keywords: Physical Therapy; low back pain,; external focus
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: 2 groups will be formed using the random randomization model
Who Masked: Participant, Outcomes Assessor
Masking Description: the participant and evaluator do not know who the groups are
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigation of the Effects of External Focused Ex. on Functionality in Individuals (Other): Sub-branches of the study are planned as Investigation of the Effects of External Focused Dynamic Balance Training on Functionality in Individuals with Chronic Low Back Pain. Sub-branches of the study are planned as Investigation of the Effects of External Focused Dynamic Balance Training on Functionality in Individuals with Chronic Low Back Pain.
  Interventions: Other: external focus task focus in addition to physiotherapy and rehabilitation exercises
- Investigation of the Effects of İnternal Focused Ex. on Functionality in Individuals (Other): Sub-branches of the study are planned as Investigation of the Effects of internal Focused Dynamic Balance Training on Functionality in Individuals with Chronic Low Back Pain. Sub-branches of the study are planned as Investigation of the Effects of İnternal Focused Dynamic Balance Training on Functionality in Individuals with Chronic Low Back Pain.
  Interventions: Other: internal focus task focus in addition to physiotherapy and rehabilitation exercises

INTERVENTIONS:
Other: external focus task focus in addition to physiotherapy and rehabilitation exercises — The first study on the external focus was made in 1998 by Wulf, Ho ¨ß, & Prinz, (1998). Focusing on the inside of the body while performing a movement is called "internal (internal focus)", focusing on the outside of the body is called "external (external focus)". Previous studies have shown that external focus is substantially more effective than internal focus in the performance of a movement.
  Other Names: ext focus
  Arms: Investigation of the Effects of External Focused Ex. on Functionality in Individuals
Other: internal focus task focus in addition to physiotherapy and rehabilitation exercises — he first study on the external focus was made in 1998 by Wulf, Ho ¨ß, & Prinz, (1998). Focusing on the inside of the body while performing a movement is called "internal (internal focus)", focusing on the outside of the body is called "external (external focus)". Previous studies have shown that external focus is substantially more effective than internal focus in the performance of a movement.
  Other Names: internal focus
  Arms: Investigation of the Effects of İnternal Focused Ex. on Functionality in Individuals

SUMMARY:
Postural control methods are impaired in people with chronic low back pain. While the person maintains balance with pain relief, fear of movement and pain increase with loss of balance. It was found that externally focused exercises are more effective than internal focus exercises in terms of motor control and motor learning. To investigate the place of externally focused balance exercises in conservative treatment of target low back pain. For this purpose, approval was obtained from the clinical research ethics committee of Kırşehir Ahi Evran University, Faculty of Medicine, with the decision numbered 2022-18/163.

DETAILED DESCRIPTION:
Focusing on the inside of the body while performing a movement is called "internal (internal focus)", focusing on the outside of the body is called "external (external focus)". Many previous studies have shown that external focus is substantially more effective than internal focus in the performance of a movement.In our randomized controlled study, there were two groups and 22 people were treated in each group. Volunteers between the ages of 18-65 who had low back pain for the last 3 months and had no musculoskeletal problems were included. Balances were evaluated with Biodex Balance Device, pain with Visual Analog Scale, performance with Physical Performance Test Battery, functional level with osvewstry disability index, posture, spinal mobility,postural endurance with spinal mouse device. 8 weeks of treatment were applied to both groups as external focus and control groups. Basically similar exercises were applied to both groups, and there were tasks in the exercises in the external focus group, and the focus were on the task other than the exercise.

The results of the study show that externally focused balance exercises are effective on dynamic balance, fall risk, stability limits, physical performance, posture, spinal mobility, and postural endurance in individuals with CLBP.

ELIGIBILITY:
Inclusion Criteria:

* Those with ongoing low back pain symptoms in the last three months (diagnosed with chronic low back pain),
* Individuals between the ages of 18-65
* Pain level 3 or more according to VAS
* Individuals who volunteer to participate in the study will be included.

Exclusion Criteria:

* Individuals with lower extremity and spine orthopedic and neurological disorders,
* Having a musculoskeletal injury in the last 9 months,
* Surgery, injection, etc. for low back pain in the last 3 months. with a history of treatment
* Those who are doing any sports activity,
* Subjects who do not cooperate well will not be included in the study. Inclusion and exclusion criteria will be the same for control group participants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-03-05 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Pain level Individuals are asked to indicate the degree of pain they have on the VAS scale numbered from 0 to 10 on a straight line, with "0" being no pain and "10" being the most severe pain. | 8 weeks
  The units included in the study are the use of VAS (Visual Analog Scale) for the presence and burden of low back pain. At the beginning and end of each start-up, the presence and effect of pain is asked and taken away. The reason for preferring these variables VAS is that they have high validity and reliability. Individuals are asked to indicate the degree of pain they have on the VAS scale numbered from 0 to 10 on a straight line, with "0" being no pain and "10" being the most severe pain.
Evaluation of Functional Status (Oswestry Disability Index) Physical functions .The result is calculated with the formula "patient's score / probable maximum score X 100". Each question has an answer rating from 0 to 5. | 8 weeks
  Oswestry Disability Scale Evaluation of Physical Function Evaluation of Functional Status (Oswestry Disability Index) Physical functions will be evaluated with the Oswestry low back pain scale. It is a very common scale compiled to evaluate the general condition of the low back in patients with low back pain. Scoring of the answered questions is carried out by adding the numbers next to the checked box. Each question has an answer rating from 0 to 5. The maximum score can be 50 if the individual has answered each question. The result is calculated with the formula "patient's score / probable maximum score X 100"
The Physical Performance Level | 8 weeks
  The physical performance test battery includes the following tests: lumbar flexion range of motion, walking fifty steps, walking for 5 minutes, sitting and standing with 5 repetitions, trunk flexion with 10 repetitions, and reaching forward with weight.
Balance | 8 weeks
  The Biodex stability system (Biodex Medical System Inc., NY, USA, Model SW4530DE6N, SD 950304) was used to assess static and dynamic balance, fall risk, and the limit of stability
Assessment of Posture, Spinal Mobility, and Postural Endurance Spinal Mobilite | 8 weeks
  Spinal posture, spinal mobility, and postural competence were measured with a computer-assisted wireless Spinal Mouse device (the Spinal Mouse System, Idiag, Fehraltorf, Switzerland). By moving the Spinal Mouse device on the spine with its wheel, it measures the length of the spine, posture, and joint movements and transfers this sequence to the computer environment. Trunk flexion posture was recorded for spinal mobility. Upright posture was measured for the postural endurance (competence) values, and then, after holding a weight of 5% of the person's body weight between the hands parallel to the shoulder level for 30 seconds, the upright posture was re-measured while the weight was still in the person's hand.

CONTACTS AND LOCATIONS:
Overall Officials: anıl özüdoğru, Principal Investigator — Kırşehir Ahi Evran University School of Physical Therapy and Rehabilitationaozudogru@hotmail.com
Locations (1):
- Kirşehir Ahi Evran Univercity, Kırşehir, Kirşehi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
ıpd Decision will be made after ipd data is collected.

REFERENCES:
- [Background] Wulf G, Lauterbach B, Toole T. The learning advantages of an external focus of attention in golf. Res Q Exerc Sport. 1999 Jun;70(2):120-6. doi: 10.1080/02701367.1999.10608029. PMID 10380243